CLINICAL TRIAL: NCT04835025
Title: A Retrospective, Multicenter Case-control Study of Radiotherapy Combined With Immunotherapy for Brain Metastases of Non-small Cell Lung Cancer
Brief Title: Radiotherapy Combined With Immunotherapy for Brain Metastases of Non-small Cell Lung Cancer
Status: Suspended | Type: Observational
Why Stopped: because of COVID-19
Sponsor: Tongji Hospital (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Wuhan University (Other); Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: TJ-IRB20210338
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Control group (radiotherapy group): In non-small cell lung cancer, patients with brain metastases received radiotherapy for brain lesion (without limitation of dose and treatment method for radiotherapy) , but not receiving immunotherapy. Those patients would enter the control group. After patients experiencing disease progression(PD) in this group, follow-up treatment does not include immunotherapy until tumor progression again or death.
  Interventions: Drug: PD-1/PD-L1 inhibitor

INTERVENTIONS:
Drug: PD-1/PD-L1 inhibitor — In non-small cell lung cancer, patients with brain metastases received radiotherapy for brain lesions and immunotherapy (including sequential and concurrent model). Those patients would enter the trial group; After patients experiencing PD in this group, follow-up treatment until tumor progression again or death

SUMMARY:
This is a Retrospective, Multicenter, Controlled Study to Evaluate Immunotherapy and Radiotherpay for Brain Lesions as a Potential Treatment for Patients with Brain Metastasis in non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

Experimental group:

1. 18 years old ≤ age ≤ 75 years old, no gender limitation;
2. NSCLC who have received radiotherapy for brain lesions + PD-1/PD-L1 immunotherapy;
3. Histologically confirmed as NSCLC;
4. Imaging confirmed brain metastasis (CT or MRI);
5. The presence of imaging-evaluable lesions can be evaluated in accordance with RECIST 1.1

Control group:

1 18 years old ≤ age ≤ 75 years old, no gender limitation; 2 NSCLC who has received radiotherapy for brain lesions; 3 Histologically confirmed as non-small cell lung cancer; 4 Imaging confirmed brain metastasis (CT or MRI); 5 The presence of imaging-evaluable lesions can be evaluated in accordance with RECIST 1.1

-

Exclusion Criteria:

1 The age is less than 18 years old, regardless of gender; 2 Histologically confirmed as NSCLC 3 Imaging confirmed the absence of brain metastases 4 NSCLC with brain metastasis only received chemotherapy or targeted therapy, and did not receive radiotherapy or immunotherapy

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. 18 years old ≤ age ≤ 75 years old, no gender limitation;
  2. NSCLC who have received radiotherapy for brain lesions ±PD-1/PD-L1 immunotherapy;
  3. Histologically confirmed as non-small cell lung cancer;
  4. Imaging confirmed brain metastasis (CT or MRI)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
progression-free surival | 3 years
  Progression-free survival: From the first treatment to the date of first documentation of disease progression, or death due to any cause

SECONDARY OUTCOMES:
overall survival | 3 years
  Overall survival: From the first administration to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, 430030, Hubei, P. R. China, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bade BC, Dela Cruz CS. Lung Cancer 2020: Epidemiology, Etiology, and Prevention. Clin Chest Med. 2020 Mar;41(1):1-24. doi: 10.1016/j.ccm.2019.10.001. PMID 32008623
- [Result] Nasim F, Sabath BF, Eapen GA. Lung Cancer. Med Clin North Am. 2019 May;103(3):463-473. doi: 10.1016/j.mcna.2018.12.006. PMID 30955514
- [Result] Rodriguez-Canales J, Parra-Cuentas E, Wistuba II. Diagnosis and Molecular Classification of Lung Cancer. Cancer Treat Res. 2016;170:25-46. doi: 10.1007/978-3-319-40389-2_2. PMID 27535388
- [Result] Wang S, Hu C, Xie F, Liu Y. Use of Programmed Death Receptor-1 and/or Programmed Death Ligand 1 Inhibitors for the Treatment of Brain Metastasis of Lung Cancer. Onco Targets Ther. 2020 Jan 23;13:667-683. doi: 10.2147/OTT.S235714. eCollection 2020. PMID 32158220
- [Result] Li W, Yu H. Separating or combining immune checkpoint inhibitors (ICIs) and radiotherapy in the treatment of NSCLC brain metastases. J Cancer Res Clin Oncol. 2020 Jan;146(1):137-152. doi: 10.1007/s00432-019-03094-9. Epub 2019 Dec 7. PMID 31813004
- [Result] Jones GS, Baldwin DR. Recent advances in the management of lung cancer. Clin Med (Lond). 2018 Apr 1;18(Suppl 2):s41-s46. doi: 10.7861/clinmedicine.18-2-s41. PMID 29700092
- [Result] Chen Y, Gao M, Huang Z, Yu J, Meng X. SBRT combined with PD-1/PD-L1 inhibitors in NSCLC treatment: a focus on the mechanisms, advances, and future challenges. J Hematol Oncol. 2020 Jul 28;13(1):105. doi: 10.1186/s13045-020-00940-z. PMID 32723363
- [Result] Qian JM, Martin AM, Martin K, Hammoudeh L, Catalano PJ, Hodi FS, Cagney DN, Haas-Kogan DA, Schoenfeld JD, Aizer AA. Response rate and local recurrence after concurrent immune checkpoint therapy and radiotherapy for non-small cell lung cancer and melanoma brain metastases. Cancer. 2020 Dec 15;126(24):5274-5282. doi: 10.1002/cncr.33196. Epub 2020 Sep 14. PMID 32926760
- [Result] Eguren-Santamaria I, Sanmamed MF, Goldberg SB, Kluger HM, Idoate MA, Lu BY, Corral J, Schalper KA, Herbst RS, Gil-Bazo I. PD-1/PD-L1 Blockers in NSCLC Brain Metastases: Challenging Paradigms and Clinical Practice. Clin Cancer Res. 2020 Aug 15;26(16):4186-4197. doi: 10.1158/1078-0432.CCR-20-0798. Epub 2020 Apr 30. PMID 32354698
- [Result] Protopapa M, Kouloulias V, Nikoloudi S, Papadimitriou C, Gogalis G, Zygogianni A. From Whole-Brain Radiotherapy to Immunotherapy: A Multidisciplinary Approach for Patients with Brain Metastases from NSCLC. J Oncol. 2019 Feb 3;2019:3267409. doi: 10.1155/2019/3267409. eCollection 2019. PMID 30853981
- [Result] Miyamoto S, Nomura R, Sato K, Awano N, Kuse N, Inomata M, Izumo T, Terada Y, Furuhata Y, Bae Y, Kunitoh H. Nivolumab and stereotactic radiation therapy for the treatment of patients with Stage IV non-small-cell lung cancer. Jpn J Clin Oncol. 2019 Feb 1;49(2):160-164. doi: 10.1093/jjco/hyy171. PMID 30452687
- [Result] Vilarino N, Bruna J, Bosch-Barrera J, Valiente M, Nadal E. Immunotherapy in NSCLC patients with brain metastases. Understanding brain tumor microenvironment and dissecting outcomes from immune checkpoint blockade in the clinic. Cancer Treat Rev. 2020 Sep;89:102067. doi: 10.1016/j.ctrv.2020.102067. Epub 2020 Jul 7. PMID 32682248
- [Result] Kowalski ES, Remick JS, Sun K, Alexander GS, Khairnar R, Morse E, Cherng HR, Berg LJ, Poirier Y, Lamichhane N, Becker S, Chen S, Molitoris JK, Kwok Y, Regine WF, Mishra MV. Immune checkpoint inhibition in patients treated with stereotactic radiation for brain metastases. Radiat Oncol. 2020 Oct 27;15(1):245. doi: 10.1186/s13014-020-01644-x. PMID 33109224